CLINICAL TRIAL: NCT03657446
Title: Randomized, Double-blind (for Clazosentan), Placebo- and Moxifloxacincontrolled, 3-way Cross-over Phase 1 Study to Assess the Effect of Two Intravenous Doses of Clazosentan on the QTc Interval Duration in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Investigate Whether Administration of Clazosentan Can Affect Normal Heart Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ID-054-107; 2018-002118-12 (EudraCT Number)
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — clazosentan; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: 3-way cross-over Phase 1 study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment sequence ABC (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacin
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin
- Treatment sequence ACB (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacinn
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin
- Treatment sequence BAC (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacin
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin
- Treatment sequence BCA (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacin
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin
- Treatment sequence CBA (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacin
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin
- Treatment sequence CAB (Experimental): Period A: clazosentan Period B: placebo Period C: placebo + moxifloxacin
  Interventions: Drug: Clazosentan; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Clazosentan — Continuous i.v. infusion of 20 mg/h or 60 mg/h of clazosentan for 3 h
Drug: Placebo — Matching placebo infusion
Drug: Moxifloxacin — Film-coated tablet containing 400 mg moxifloxacin

SUMMARY:
The study will investigate whether administration of clazosentan can affect normal heart function in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

General criteria

* Signed informed consent prior to any study-mandated procedure
* Body mass index of 18.0-30.0 kg/m2 (inclusive) at Screening
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on the same arm, after 5 min in the supine position at Screening and on Day -1 of the first Period
* 12-lead ECG: QT interval corrected using Fridericia's formula (QTcF) <450 ms for male subjects and < 470 ms for female subjects, QRS interval < 110 ms, PR interval ≤ 200 ms, and heart rate (HR) ≤ 90 bpm without clinically relevant abnormalities using a 12-lead ECG measured after 5 min in the supine position at Screening and on Day -1 of the first Period

Study-specific criteria

* Women of non-childbearing potential
* Male subjects must accept to use a condom and not to procreate for the duration of the study and for 3 months thereafter

Exclusion Criteria:

General criteria

* Previous exposure to clazosentan or to moxifloxacin within 3 months prior to Screening
* Known hypersensitivity to any of clazosentan excipients or to moxifloxacin or any of its excipients
* Any contraindication to moxifloxacin treatment
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the study
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions if considered clinically significant by the investigator
* Veins unsuitable for i.v. puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture)
* Participation in a clinical study involving study treatment administration within 3 months prior to Screening or in more than 4 clinical studies within 1 year prior to Screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Study-specific criteria

• History or presence of rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change-from-baseline QTcF (ΔΔQTcF) with its upper limit of the two-sided 95% confidence interval (CI) | From 1 hour pre-dose to 24 hour after the end of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrich A, Juif PE, Dingemanse J, Krause A. PK/PD modeling of a clazosentan thorough QT study with hysteresis in concentration-QT and RR-QT. J Pharmacokinet Pharmacodyn. 2021 Apr;48(2):213-224. doi: 10.1007/s10928-020-09728-7. Epub 2021 Jan 2. PMID 33389549